CLINICAL TRIAL: NCT07336251
Title: Transcranial Magnetic Stimulation in Veterans With PTSD: A Pilot Study to Examine Mechanism of Effect
Brief Title: Transcranial Magnetic Stimulation in Veterans With PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bradley Watts, Staff Psychiatrist, White River Junction Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1869595
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: PTSD - Post Traumatic Stress Disorder
MeSH Terms: conditions — Combat Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants receiving open label trial of TMS (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — 10 sessions of low frequency rTMS (1Hz) applied to the right dorsolateral prefrontal cortex.

SUMMARY:
With this research investigators hope to begin to understand how rTMS can improve posttraumatic stress disorder (PTSD) symptoms. TMS improves PTSD through two interrelated mechanisms: change in brain limbic system function and change in systemic inflammatory activation. Participants who decide to join this study, will receive ten rTMS treatments. All participants will undergo a 40-minute rTMS procedure with a member of the study team 10 times over 2-4 weeks. Participants will undergo fMRI scans of the head in order to help researchers better understand potential effects of rTMS on brain activity. In addition, participants will be asked to give two breath and blood samples to look for signs of general inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 70
* Eligible for VA healthcare
* Moderate to severe PTSD as determined by a total score of at least 25 on the CAPS within 7 days of randomization.
* Agree to have CAPS audio recorded.
* Ability to obtain a Motor Threshold using the TMS device during screening.
* If female with childbearing potential, use of acceptable method of birth control (i.e., use of contraceptives, abstinence).
* Able to read, understand, and sign the informed consent document.

Exclusion Criteria:

* Pregnant or lactating woman.
* MRI is contraindicated
* Current use of clozapine (any dose) or bupropion (more than 300mg per day).
* Cardiac pacemaker or implantable defibrillator.
* Presence of any metal object in the head, including cochlear implants, but excluding dental work in the mouth.
* Significant central nervous system disorder (stroke, brain mass, epilepsy).
* Seizure in past one year.
* Current psychosis or mania.
* Significant suicidal ideation.
* Unstable medical conditions.
* Current alcohol or substance use disorder (except nicotine) that interferes with the patient's ability to participate.
* CPT or PE for PTSD in the past 2 months.
* Changes in Fluoxetine, Paroxetine, Sertraline, or Venlafaxine in the past 2 months.
* Color blind
* Currently participating in other research studies.
* Aneurysm Clip
* Ocular foreign body (e.g., metal shavings)
* Any implanted device (pumps, infusion devices, etc.)
* Shrapnel injuries or metal fragments

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and intensity of PTSD symptoms as assessed by the CAPS-5 | From enrollment to the end of treatment at 3 months
  The CAPS is a clinician-administered scale of PTSD symptoms, which queries the frequency and intensity of symptoms of PTSD
20 item self-report of PTSD symptoms assessed by PCL-5 | From enrollment to the end of treatment at 3 months
  It asks participants to rate the severity of each of the 20 symptoms of PTSD in DSM-5

SECONDARY OUTCOMES:
A quick self-reported and self administered inventory of depressive symptoms (QIDS-16-SR) | From the baseline to the end of the study at 3 months
  This is a self-reported, self- administered scale of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Watts, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- White River Junction VA Hospital, White River Junction, Vermont, United States